CLINICAL TRIAL: NCT06373172
Title: Enhancing Clinical Reasoning Competency for Undergraduate Nursing Students Using Virtual Simulation-based Education Based on the Rasch Model
Brief Title: Enhancing Clinical Reasoning Competency
Acronym: Reasoning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongmyong University (Other)
Responsible Party: Principal Investigator, Sung Hae Kim, Assistant professor, Tongmyong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202005-HR-003
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Clinical Reasoning; Communication; Development, Human
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This quasi-experimental study used a single-group pretest-posttest design to verify the effectiveness of virtual simulation-based education for undergraduate nursing students.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhancing Clinical Reasoning Competency for Undergraduate Nursing Students (Experimental): Enhancing Clinical Reasoning Competency for Undergraduate Nursing Students Using Virtual Simulation-based Education based on the Rasch model
  Interventions: Other: virtual simulation-based education program

INTERVENTIONS:
Other: virtual simulation-based education program — We used "vSim® for Nursing - Nursing Medical-Surgical" as the virtual simulation-based education program. Four modules were included: (a) acute myocardial infarction, (b) diabetes mellitus, (c) transfusion, and (4) asthma. Each module learning sessions was conducted based on scenarios, which consisted of five steps: Suggested reading, Pre-simulation quiz, vSim, Post-simulation quiz, and Guide reflection questions. For each module, the intervention was performed for two hours. The participants attended four module learning sessions and received eight hours of training. Debriefing using guided reflection questions were completed in the form of a team reflection, followed by an instructor-learner discussion and feedback for 20 minutes of each module.

SUMMARY:
Enhancing Clinical Reasoning Competency for Undergraduate Nursing Students Using Virtual Simulation-based Education based on the Rasch model

Aims: Clinical reasoning is a core nursing competency that involves analyzing patient-related data and providing appropriate nursing practices. Simulation-based education is effective in improving the clinical reasoning competencies and communication skills of nursing students. This study aimed to verify the effectiveness of virtual simulation-based education.

DETAILED DESCRIPTION:
Methods: This study used a single-group pre- and post-test experimental design to verify the effectiveness of virtual simulation-based education. Data were collected from June to September 2020. Thirty-six nursing students in the 3rd and 4th grades who understood the purpose of this study were selected as participants. The collected data were analyzed using SPSS Statistics 25.0 and Winsteps 3.68.2.

Keywords: Clinical Reasoning, Competency, Communication, Nursing, Virtual Simulation

ELIGIBILITY:
Inclusion Criteria:

* The participants were third- and fourth-year undergraduate nursing students who understood the purpose of the study and voluntarily agreed to participate

Exclusion Criteria:

* A person who has difficulty communicating or has no willingness to participate

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Nurses Clinical Reasoning Scale | 4month
  The Nurses Clinical Reasoning Scale (NCRS) includes 15 items rated on a five-point Likert scale (1=Strongly disagree, 5=Strongly agree, min:15 & max:75) (Liou et al., 2016). We used the Korean version of the NCRS in this study (Joung & Han, 2017). Higher scores indicated better clinical reasoning. Cronbach's α was 0.94 for the original NCRS, and 0.93 for the Korean version of the NCRS.
Communication Skills Scale | 4month
  The Global Interpersonal Communication Competence Scale (GICC-15) includes 15 items rated on a five-point Likert scale (1= strongly disagree to 5= strongly agree. min:15 & max:75) (Rubin & Martin, 1994). We used the Korean version of the GICC-15 (Hur, 2003). Cronbach's α in Hur's (2003) study was 0.72.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hae Kim, PhD, Principal Investigator — Tongmyong University
Locations (1):
- Tongmyong Unoversity, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No